CLINICAL TRIAL: NCT03907111
Title: Develop the Biologic-fibrotic Dressing on War Open Bleeding Wounds for Hemostasis.
Brief Title: Compare the Hemostatic Effectiveness of Chitosan Gauze With Traditional Gauze on Open Wound on 10 Participants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Hsu Sheng-Der, attending physician, department of traumatology, Tri-Service General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hemostatic-Chitosan-2015
Record Dates: First submitted 2019-04-03; First posted 2019-04-08 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Hemostasis
Keywords: bleeding wounds, hemostasis, open wounds, infection, antimicrobial
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Each of the participants was been treated with 2 different treatments on different areas of the same wound at the same time.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chitosan gauze (Experimental): 100cm^2 Gauze made by chitosan material. Administrate it on surgical wound after surgery directly. Change it daily with necessary wound care.
  Interventions: Device: Chitosan Gauze
- Traditional gauze (Placebo Comparator): 100cm^2 Gauze made by traditional cotton yarn. Administrate it on surgical wound after surgery directly. Change it daily with necessary wound care.
  Interventions: Device: placebo

INTERVENTIONS:
Device: Chitosan Gauze — Gauze made by chitosan material
  Arms: Chitosan gauze
Device: placebo — traditional gauze
  Arms: Traditional gauze

SUMMARY:
This study recruited 10 subject participants to compare the hemostasis gauze made by chitosan with traditional cotton gauze to see which one is better in bleeding time, bleeding volume, wound infection and wound healing speed when it is used in open wound treatment.

DETAILED DESCRIPTION:
open wound bleeding and infection care policy development is focusing on efficiency to strengthen internal bleeding, pain, avoidance of infection and promoting wound healing wound. With the changes in the social environment, people caring for hemostasis and wound healing have become increasingly demanding. Presently, studies generally aim to stop the bleeding using trauma care technology and functional capabilities combined with each other as well as inhibit lower infection and can also help assist healing wounds care strategy for the protection of human lives. Therefore, the goal of the plan is to establish new care strategies on open wounds infection to stop the bleeding and to improve the health and safety of the people. The researchers will choose the general biological hemostatic gauze to conduct clinical trials comparing the clinical hemostasis focusing on bleeding time, wound infection in the wound and the wound bacteria penetrating situations in the hope to build a better strategy in rapid hemostasis and wound infection care strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patients need laparotomy, with the expected wound size bigger than 5 cm in length and 2 cm in width.

Exclusion Criteria:

* Have history of allergy to shrimp, crab and other chitins.
* Patients with blood clotting disorders
* Vulnerable group
* Patients with unstable vital sign

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-10-02 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-02-10 (Actual)

PRIMARY OUTCOMES:
Time to Hemostasis | one hour after the surgery
  How many second it takes to stop bleeding

SECONDARY OUTCOMES:
Breeding volume | one hour after the surgery
  the weight gain of the gauze from it been administrated on the wound until the hemostasis of the wound.
Relative light units difference | day0, day7 and day 14.
  compare the relative light unit(RLU, relative light units, is by detecting the ATP concentration in the samples to determine the relative bacteria number, kikkoman PD-30) difference on the gauze collected at the daily wound care between chitosan gauze and traditional gauze.
size of the wound in millimeter | day1, day3, day 5, day7 and day14.
  observe the difference of size between different treatment.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hattori H, Amano Y, Nogami Y, Takase B, Ishihara M. Hemostasis for severe hemorrhage with photocrosslinkable chitosan hydrogel and calcium alginate. Ann Biomed Eng. 2010 Dec;38(12):3724-32. doi: 10.1007/s10439-010-0121-4. Epub 2010 Jul 9. PMID 20617383
- [Background] Charlesworth TM, Agthe P, Moores A, Anderson DM. The use of haemostatic gelatin sponges in veterinary surgery. J Small Anim Pract. 2012 Jan;53(1):51-6. doi: 10.1111/j.1748-5827.2011.01162.x. PMID 22212190
- [Background] Goyal AK, Garg T, Rath G, Gupta UD, Gupta P. Development and Characterization of Nanoembedded Microparticles for Pulmonary Delivery of Antitubercular Drugs against Experimental Tuberculosis. Mol Pharm. 2015 Nov 2;12(11):3839-50. doi: 10.1021/acs.molpharmaceut.5b00016. Epub 2015 Oct 5. PMID 26436948
- [Background] Bozkir A, Saka OM. Chitosan-DNA nanoparticles: effect on DNA integrity, bacterial transformation and transfection efficiency. J Drug Target. 2004 Jun;12(5):281-8. doi: 10.1080/10611860410001714162. PMID 15512779
- [Background] Wang CC, Su CH, Chen CC. Water absorbing and antibacterial properties of N-isopropyl acrylamide grafted and collagen/chitosan immobilized polypropylene nonwoven fabric and its application on wound healing enhancement. J Biomed Mater Res A. 2008 Mar 15;84(4):1006-17. doi: 10.1002/jbm.a.31482. PMID 17647243
- [Background] Koca Kutlu A, Cecen D, Gurgen SG, Sayin O, Cetin F. A Comparison Study of Growth Factor Expression following Treatment with Transcutaneous Electrical Nerve Stimulation, Saline Solution, Povidone-Iodine, and Lavender Oil in Wounds Healing. Evid Based Complement Alternat Med. 2013;2013:361832. doi: 10.1155/2013/361832. Epub 2013 Jun 3. PMID 23861704
- [Background] Kordjazi M, Shabanpour B, Zabihi E, Faramarzi MA, Feizi F, Ahmadi Gavlighi H, Feghhi MA, Hosseini SA. Sulfated polysaccharides purified from two species of padina improve collagen and epidermis formation in the rat. Int J Mol Cell Med. 2013 Fall;2(4):156-63. PMID 24551807
- [Background] Junker JP, Kamel RA, Caterson EJ, Eriksson E. Clinical Impact Upon Wound Healing and Inflammation in Moist, Wet, and Dry Environments. Adv Wound Care (New Rochelle). 2013 Sep;2(7):348-356. doi: 10.1089/wound.2012.0412. PMID 24587972